CLINICAL TRIAL: NCT07025486
Title: Effectiveness of HabitWorks and Symptom Tracking for Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Courtney Beard, PhD, Associate Professor, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P001752
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Depression, Anxiety
Keywords: interpretation bias; digital mental health
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HabitWorks + Symptom Tracking (Experimental): Use of HabitWorks app 3 times/week for 4 weeks + weekly symptom tracking
  Interventions: Behavioral: HabitWorks; Behavioral: Symptom TRacking
- Symptom Tracking (Active Comparator): Symptom Tracking 3 times per week for 4 weeks
  Interventions: Behavioral: Symptom TRacking

INTERVENTIONS:
Behavioral: HabitWorks — Smartphone delivered interpretation bias exercises, symptom tracking
  Arms: HabitWorks + Symptom Tracking
Behavioral: Symptom TRacking — Self-assessment via symptom surveys

SUMMARY:
Our objective is to conduct a randomized controlled trial (RCT) that compares two digital interventions - Symptom Tracking and the HabitWorks app - in a sample of adults endorsing symptoms of anxiety or depression. We hope to obtain pilot data to support a fully powered RCT to test moderators:

1. Target engagement (improvement in interpretation bias)
2. Feasibility and acceptability of Symptom Tracking and HabitWorks and procedures for a general community sample
3. Symptom and functioning measures

DETAILED DESCRIPTION:
HabitWorks is a personalized, transdiagnostic, smartphone-delivered interpretation bias intervention. Our pilot studies of HabitWorks revealed good acceptability, feasibility, and target engagement in a variety of populations (Beard, Ramadurai, et al., 2021; Beard, Beckham, et al., 2021). Our next step is to test effectiveness for anxiety and depression symptoms in a larger, community sample. Results will provide pilot data to support an R01 effectiveness trial. We will randomize adults with anxiety or depression to HabitWorks or a credible control arm and examine effects on interpretation bias, symptoms, and functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 at the time of consent (19 in Nebraska, 21 in Puerto Rico based on age of consent)
2. Current US resident
3. Total score ≥ 3 on the Patient Health Questionnaire-2 (Kroenke et al., 2003) or Generalized Anxiety Disorder-2 (Spitzer et al., 2006), indicating at least mild depression and/or anxiety symptoms
4. 24-hour access to an iPhone smartphone
5. ability to understand English

Exclusion criteria:

1. No current psychiatric symptoms that would prevent informed consent, understanding of research procedures, or ability to complete the study (e.g., active symptoms of psychosis, mania)
2. No medical symptoms that would prevent informed consent, understanding of research procedures, or ability to complete the study (e.g., physical disability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
GAD-7 | From enrollment to the end of followup period at 8 weeks
  self-report measure of general anxiety symptoms, completed online via RedCap

SECONDARY OUTCOMES:
Clinical Global Improvement Scale | post-treatment (4 weeks after enrollment)
  self-reported single item assessing perceived improvement due to a treatment

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
STudy protocol, statistical plan, analytic code will be shared on open science framework
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: anticipated July 2025 with no end date
Access Criteria: open science framework